CLINICAL TRIAL: NCT02331979
Title: Improving Bladder Function in SCI by Neuromodulation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Daniel Lu, MD, PhD, Associate Professor, University of California, Los Angeles
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14-000932
Record Dates: First submitted 2015-01-03; First posted 2015-01-06 (Estimated); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Spinal Cord Injury
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Stimulation of Non-Naive (Experimental): Evaluate neuromodulation in 6 subjects with prior motor training.
  Interventions: Device: Electromagnetic Neuromodulation
- Stimulation of Naive (Experimental): Evaluate neuromodulation in 6 naive subjects.
  Interventions: Device: Electromagnetic Neuromodulation
- Stimulation (Experimental): Apply parameters discovered in Arm 1 and Arm 2 to evaluate neuromodulation in 12 naive subjects.
  Interventions: Device: Electromagnetic Neuromodulation

INTERVENTIONS:
Device: Electromagnetic Neuromodulation — Electromagnetic stimulation to neuromodulate the spinal cord in the context of spinal cord injury.
  Other Names: Transcutaneous Electrical Stimulation; Magnetic Stimulation

SUMMARY:
This trial will investigate the safety and utility of spinal cord neuromodulation to improve urinary bladder function in the context of spinal cord injury.

DETAILED DESCRIPTION:
This trial will investigate the safety and utility of spinal cord neuromodulation to improve urinary bladder function in the context of spinal cord injury. Neuromodulation will be in the form of transcutaneous electrical stimulation and/or magnetic stimulation.

ELIGIBILITY:
Inclusion Criteria:

1. Male 18-45 years;
2. At least 1 year post-injury;
3. Non-progressive SCI at C2-T8 (non-conus injury);
4. Motor Complete ASIA (A or B);
5. Neurogenic bladder requiring clean intermittent straight catheterization;
6. Able to attend twice weekly testing sessions for 6 months.
7. Have intact lower extremity anatomy and able to use lower extremity for assistive standing and stepping.

Exclusion Criteria:

1. History of autonomic dysreflexia;
2. Ventilator dependency;
3. Musculoskeletal dysfunction, unhealed fracture, pressure ulcer, active infection;
4. Clinically significant depression or ongoing drug abuse;
5. Received botox injection, or bladder surgery (suprapubic access, Brindley procedure, etc.); 6. Prostatic hypertrophy or bladder outlet disorder;

7. Cardiopulmonary disease that precludes lower extremity training or rehabilitation.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2015-09; Primary Completion 2025-12-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Urine flow and volume | Months 1-48

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States